CLINICAL TRIAL: NCT04516070
Title: Stereotactic Radiosurgery (SRS) as Definitive Management for a Limited Number of Small Cell Lung Cancer (SCLC) Brain Metastasis
Brief Title: Stereotactic Radiosurgery for the Treatment of Patients With Small Cell Lung Cancer Brain Metastasis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0900; NCI-2020-05720 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0900 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Lung Small Cell Carcinoma; Metastatic Malignant Neoplasm in the Brain; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Small Cell Lung Carcinoma; Brain Neoplasms; Lung Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (SRS) (Experimental): Patients undergo SRS in the absence of disease progression or unacceptable toxicity. Patients whose disease progresses may be treated with additional courses of SRS per physician discretion.
  Interventions: Other: Questionnaire Administration; Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Radiosurgery — Undergo SRS
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery

SUMMARY:
This phase II trial investigates how stereotactic radiosurgery affects brain functions while treating patients with small cell lung cancer that has spread to the brain (brain metastasis). Standard of care treatment consists of whole brain radiation therapy, which targets the entire brain, and may result in side effects affecting the nervous system. Stereotactic radiosurgery only targets areas of the brain that are suspected to be affected by the disease. The purpose of this trial is to learn if and how patients' brain functions are affected by the use of stereotactic radiosurgery rather than whole brain radiation therapy in managing brain metastasis caused by small cell lung cancer. Stereotactic radiosurgery may help patients avoid nervous system side effects caused by whole brain radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the cognitive decline rate at 3 months.

SECONDARY OBJECTIVES:

I. To examine cognitive decline rate on each individual cognitive test at each time point.

II. To examine cognitive decline rates using reliable change index methodology. III. To report the overall survival of patients (death due to any cause) of patients receiving stereotactic radiosurgery (SRS) for small cell lung cancer (SCLC) brain metastasis.

IV. To report rates of local tumor control (of the treated lesions) in the brain post-treatment, as dictated by magnetic resonance imaging (MRI) surveillance schedule above.

V. To report distant tumor control in the brain (of non-treated lesions) post-treatment, as dictated by MRI surveillance schedule above.

VI. To report time elapsed from SRS to whole brain radiation therapy (WBRT). VII. To report rate of intracranial toxicity of SRS in the setting of prior WBRT.

VIII. To report rates of intracranial toxicity of concurrent atezolizumab with SRS.

IX. To determine rates of systemic and intracranial disease control (time to progression) in those who are treated concurrently with atezolizumab and SRS.

X. To determine the rates of SCLC-specific survival. XI. To assess the pre-treatment factors and baseline characteristics in the predictive determination of local control, intracranial control, systemic control, and neurocognitive outcomes.

XII. To assess the correlation between number of lesions and total volume of intracranial disease and neurocognitive outcome.

XIII. To document post-treatment intracranial toxicity profile in patients after SRS.

CORRELATIVE OBJECTIVE:

I. Cerebral spinal fluid (CSF) biomarkers.

OUTLINE:

Patients undergo SRS in the absence of disease progression or unacceptable toxicity. Patients whose disease progresses may be treated with additional courses of SRS per physician discretion.

After completion of study treatment, patients are followed up at 1, 3, 6, 9, 12, 16, 20, 24, 30, and 36 months after SRS.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have Eastern Cooperative Oncology Group (ECOG) =< 3
* All patients must have histologic evidence suggesting small cell lung cancer. Histologic confirmation may be from the primary tumor site, or from another metastatic site (systemic lymph node, etc.). Cytology-alone is not an acceptable method of diagnosis.
* Patient has 10 or less brain metastases on contrast-enhanced brain MRI scan obtained no greater than 6 weeks prior to study registration. Biopsy of brain metastasis is not required. A patient may be enrolled with zero brain metastasis assuming that the SRS is to be directed at the post-operative surgical cavity of a resected metastasis.
* Patients must be eligible to have all lesions treated with stereotactic radiosurgery as determined by the study radiation oncologist
* Patients must sign informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of the hospital
* Patients should have normal coagulation [International Normalized Ratio (INR) < 1.3]. within 28 days of enrollment.
* Patient's primary language is English
* No prior radiation therapy to the brain, including WBRT, PCI, or SRS
* Performance Status Assessment
* Standard ECOG performance status assessment will be used and determined by the treating physician

Exclusion Criteria:

* Patients are excluded if they have a history of metastatic cancer in addition to small cell malignancy or a history of uncontrolled non-metastatic cancer. Patients with localized squamous cell carcinoma and/or basal cell carcinoma are not excluded
* Patients are excluded if there is radiographic evidence of leptomeningeal disease
* Patients are excluded if there are malignant cells identified in the CSF on cytologic examination
* Patients are not excluded for circulating tumor deoxyribonucleic acid (DNA) (ctDNA) found in the CSF
* Female patients of childbearing age are excluded if they are pregnant as determined with a urine or serum beta human chorionic gonadotropin (HCG) no greater than 14 days prior to study registration, or breast-feeding
* Patients are excluded if they are unable to obtain an MRI scan for any other reason, including gadolinium allergy
* Patients are excluded with medical history of a psychiatric or neurologic illness, or other comorbidities believed to affect cognitive function. Subjects with neurocognitive deficit related to brain metastasis are an exception to this criterion and may qualify for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive decline | At 3 months post-stereotactic radiosurgery (SRS)
  Will be defined as a decline of >= 1 standard deviation from baseline on at least 1 of the 5 cognitive tests. Will be estimated along with the 95% confidence interval. For patients with or without prior radiation therapy to the central nervous system, the cognitive decline rate will also be estimated respectively. Fisher exact test will be used to compare the neurocognitive decline rate at 3 month post-SRS in subgroups (e.g. prior therapy difference).
Incidence of adverse events | Up to 36 months
  All toxicities will be assessed with National Cancer Institute predefined Common Terminology Criteria for Adverse Events version 5.

SECONDARY OUTCOMES:
Cognitive decline | Up to 36 months
  Will use descriptive statistics and boxplots to summarize and illustrate the neurocognitive function score at each assessment time.
Change in neurocognitive score | Baseline, up to 36 months
  Will summarize and illustrate the change from baseline in neurocognitive score. Will also model the cognitive data with mixed effects regression including baseline neurocognitive scores, time, and number of lesions, extra-cranial disease, and a patient specific random effect.
Overall survival | Time from SRS until death or last follow-up, assessed up to 36 months
  Will be estimated using the product-limit estimator of Kaplan and Meier, and log-rank test will be used for comparison of neurocognitive decline rate in subgroups (e.g. prior radiation treatment status). Cox proportional hazards regression will be used to model time to event survival as a function of age, performance status, extra-cranial disease, and other factors.
Small cell lung cancer (SCLC)-specific survival | Time from SRS till SCLC-related death or last follow-up, assessed up to 36 months
  Will be estimated using the product-limit estimator of Kaplan and Meier, and log-rank test will be used for comparison of neurocognitive decline rate in subgroups (e.g. prior radiation treatment status). Cox proportional hazards regression will be used to model time to event survival as a function of age, performance status, extra-cranial disease, and other factors.
Time to neurocognitive decline | Time from date of SRS till the cognitive decline, assessed up to 36 months
  Will be estimated using the product-limit estimator of Kaplan and Meier, and log-rank test will be used for comparison of neurocognitive decline rate in subgroups (e.g. prior radiation treatment status). Cox proportional hazards regression will be used to model time to event survival as a function of age, performance status, extra-cranial disease, and other factors.
Time duration from SRS to whole brain radiation therapy (WBRT) | Time from SRS to the start of WBRT treatment, assessed up to 36 months
  Will be estimated using the product-limit estimator of Kaplan and Meier, and log-rank test will be used for comparison of neurocognitive decline rate in subgroups (e.g. prior radiation treatment status). Cox proportional hazards regression will be used to model time to event survival as a function of age, performance status, extra-cranial disease, and other factors.
Local tumor control rates | Up to 36 months
  Will be estimated along with 95% confidence intervals. The association between the control rate and patient characteristics including pre-treatment factors (e.g. number of lesions) will be evaluated using Wilcoxon rank sum test or Fisher exact test. Logistic regression will be used to assess different patient clinical factor effect on the control rate.
Distant tumor control rate | Up to 36 months
  Will be estimated along with 95% confidence intervals. The association between the control rate and patient characteristics including pre-treatment factors (e.g. number of lesions) will be evaluated using Wilcoxon rank sum test or Fisher exact test. Logistic regression will be used to assess different patient clinical factor effect on the control rate.
Rate of systemic and intracranial disease control rate | Up to 36 months
  Will be estimated along with 95% confidence intervals. The association between the control rate and patient characteristics including pre-treatment factors (e.g. number of lesions) will be evaluated using Wilcoxon rank sum test or Fisher exact test. Logistic regression will be used to assess different patient clinical factor effect on the control rate.
Response to SRS therapy | Up to 36 months
  Will be determined by the radiology report. Will be estimated along with 95% confidence intervals. The association between the control rate and patient characteristics including pre-treatment factors (e.g. number of lesions) will be evaluated using Wilcoxon rank sum test or Fisher exact test. Logistic regression will be used to assess different patient clinical factor effect on the control rate.
Post-treatment intracranial toxicity profile | Up to 36 months
  Will be summarized and documented.
Rate of intracranial toxicity of SRS in the setting of prior WBRT | Up to 36 months
  Will be summarized according to intensity and treatment relationship, and categorized by System Organ Class.
Rate of intracranial toxicity concurrent atezolizumab with SRS | Up to 36 months
  Will be summarized according to intensity and treatment relationship, and categorized by System Organ Class.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/70/NCT04516070/ICF_000.pdf